CLINICAL TRIAL: NCT03191890
Title: Observational, Non-Interventional, Prospective, Post Market Surveillance & Post Market Clinical Follow up, International, Medical Registry to Confirm the Safety and the Performance of the Anecova Intra Uterine Culture Device for Participants With Subfertility Issue Undergoing Assisted Reproductive Medical Treatment in Routine Clinical Practice
Brief Title: Post Market Surveillance & Post Market Clinical Follow up, International, Medical Registry to Confirm the Safety and the Performance of the Anecova Intra Uterine Culture Device
Status: Withdrawn | Type: Observational
Why Stopped: Sponsor stopped the study due to poor enrollment
Sponsor: Anecova SA (Industry)
Responsible Party: Sponsor
Other Study IDs: NCV_REG_01
Record Dates: First submitted 2017-06-16; First posted 2017-06-19 (Actual); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Infertility; Reproductive Sterility
Keywords: in vivo culture
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 9 Weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is designed to generate a comprehensive survey of the use on the market of the Anecova device within its intended indications according to the Instructions For Use. The Anecova Registry is part of the Anecova quality system, to enable the Post Marketing Surveillance and the Post Market Clinical Follow-up.

DETAILED DESCRIPTION:
As soon as the very first minute of the fertilization process, very important biological events, critical for the future developmental competency of the embryo are taking place.

These biological events, after the sperm cell entry in the oocyte cytoplasm and prior to the first cleavage, include: the completion of the meiosis, the exclusion of the second polar body, the pronuclei formation, the replication of the male and female DNA and the chromosome segregation on the newly formed mitotic spindle.

If any of these events is aberrant, one or both of the two daughter cells and their descendants may carry chromosomal anomalies. In other words an uneven first cleavage in size or in content is associated with chromosomal abnormality and aneuploidy.

In vivo all these events occur in a natural environment where the presence of specific molecules and of a dynamic and physiological environment might be an advantage over in vitro culture conditions to ensure optimal cellular functions.

The Registry will capture information from the Anecova procedure, from the outcomes, from the procedure performance, from the safety and from the utilization of the Anecova Medical Device in clinical routine.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 43,
* Hormonal serum levels within normal ranges for the routinely or specifically tested hormones (FSH, LH, AMH, E2, PRL, P4, TSH),
* BMI between 18 and 29, If assessed normal antral follicular count and regular menses

Exclusion Criteria:

* Endometrial, autoimmune or hormonal specificities, as well as presence of pathology that could be potentially deleterious to the healthy development of embryos in the uterine cavity (i.e. severe endometriosis),
* Acute or chronic gynecological infection

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants following a normal course of in vitro fertilization (IVF) or intracytoplasmic sperm injection (ICSI) can benefit from the use of the Anecova device
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-06-15 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
Fertilization rate | 1 day
  Number of zygotes over all transferred injected/inseminated oocytes

SECONDARY OUTCOMES:
Biochemical Pregnancy rate | 15 days
  hCG test
Implantation rate | 5 weeks
  number of gestational sac per transferred embryos
Clinical pregnancy rate | 9 weeks
  beating heart

CONTACTS AND LOCATIONS:
Locations (1):
- IVI Bilbao, Leioa, Basque Country, Spain

IPD SHARING:
Plan to Share IPD: Undecided